CLINICAL TRIAL: NCT07382830
Title: Efficacy of Laser Pointer-Guided Visual Feedback Stabilization Exercise Program After Lumbar Microdiscectomy Surgery: A Randomized Controlled Trial
Brief Title: Effectiveness of a Visual Feedback Exercise Program Following Lumbar Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, İsmet Tümtürk, Physical therapist, MSc, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Laser Pointer Exercise
Record Dates: First submitted 2026-01-17; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Lumbar Microdiscectomy; Postoperative Rehabilitation; Randomized Controlled Trial
MeSH Terms: interventions — Exercise; Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser-Guided Exercise Group (Experimental): Participants received a supervised stabilization exercise program guided by visual feedback using a laser pointer, in addition to standard postoperative care following lumbar microdiscectomy surgery.
  Interventions: Other: Exercise
- Control Group (Active Comparator): Participants received a supervised stabilization exercise program without standard postoperative care, back training, or visual feedback following lumbar microdiscectomy surgery.
  Interventions: Other: Control

INTERVENTIONS:
Other: Exercise — Participants undergo supervised stabilization exercises for a total of 24 sessions over 8 weeks, starting 6 weeks after lumbar microdiscectomy surgery, 3 days a week. The exercises will be performed with visual feedback provided by a laser pointer placed on the lumbar region. Participants will be asked to keep the laser pointer fixed on a designated point or line on the reference diagram in front of them during the exercises. The program includes posterior pelvic tilt, partial sit-ups, bird-dog, abdominal bracing in the supine position (progression with limb movements), straight and side planks, bridge building, pelvic floor, and diaphragmatic breathing exercises. Repetitive exercises will be performed in 3 sets of 10 repetitions, while plank exercises will initially be performed in 3 repetitions of 15-30 seconds, with progression based on the individual's performance and weeks. All participants will be provided with a post-operative training program in video format.
  Other Names: Laser-Guided Supervised Exercise
  Arms: Laser-Guided Exercise Group
Other: Control — Starting 6 weeks after surgery, a supervised stabilization exercise program consisting of 24 sessions over 8 weeks, 3 days a week, will be implemented. The same exercises as in the laser group will be performed, but without the use of visual feedback. All participants will be provided with a post-operative training program in video format.
  Other Names: Control Group
  Arms: Control Group

SUMMARY:
The aim of this study is to compare the effectiveness of stabilization exercises performed with visual feedback guided by a laser pointer after lumbar microdiscectomy surgery with that of standard stabilization exercises. The study, planned as a randomized controlled trial, will include 42 individuals aged 18-65 who have undergone lumbar microdiscectomy. Participants will be divided into two groups: a control group and a laser-guided exercise group. Both groups will undergo supervised stabilization exercises 3 days a week for 8 weeks, starting from the 6th postoperative week. The outcome measures were defined as pain, disability, back awareness, trunk muscle endurance, reaction time, balance, function, and lumbar proprioception. The findings are expected to demonstrate the effectiveness of visual feedback-assisted stabilization exercises in postoperative rehabilitation and contribute to clinical practice.

DETAILED DESCRIPTION:
This study is a randomized controlled trial designed to compare the effects of stabilization exercises performed with laser-guided visual feedback and conventional stabilization exercises in individuals who have undergone lumbar microdiscectomy surgery. A total of 42 participants aged 18-65 years who have undergone lumbar microdiscectomy will be included in the study. Participants will be randomly assigned to either a control group or a laser-guided exercise group. Both groups will receive supervised stabilization exercise programs three times per week for eight weeks, starting from the sixth postoperative week. The exercise content will be similar in both groups, with the laser-guided group receiving additional visual feedback during exercises. Outcome measures will be assessed at baseline and after completion of the intervention. Assessments will include pain, disability, back awareness, trunk muscle endurance, reaction time, balance, functional performance, and lumbar proprioception. The results of this study are expected to contribute to evidence-based postoperative rehabilitation approaches following lumbar microdiscectomy.

ELIGIBILITY:
Inclusion Criteria:

* To be between 18 and 65 years of age
* Patients who underwent lumbar microdiscectomy surgery
* Individuals who are literate in Turkish

Exclusion Criteria:

* Patients who have previously undergone lumbar disc herniation surgery
* The surgical procedure involving fusion has been performed.
* Having a body mass index above 30
* Suspected or confirmed tumors in the lumbar spine and spinal canal
* Severe heart failure and cerebrovascular accident
* The presence of cauda equina syndrome and concomitant diseases of the lumbar spine
* The presence of heart conditions, orthopedic contraindications, or systemic diseases that could prevent participation in the exercise program
* Refusing to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain Assessment | All primary and secondary outcomes will be assessed at baseline (postoperative week 6) and post-intervention (postoperative week 14).
  It will be assessed using the Numerical Rating Scale (NRS).
Disability Assessment | All primary and secondary outcomes will be assessed at baseline (postoperative week 6) and post-intervention (postoperative week 14).
  It will be measured using the Oswestry Disability Index (ODI).
Lumbar Proprioception Assessment | All primary and secondary outcomes will be assessed at baseline (postoperative week 6) and post-intervention (postoperative week 14).
  It will be measured using a smartphone-based inclinometer application.
Back Awareness Assessment | All primary and secondary outcomes will be assessed at baseline (postoperative week 6) and post-intervention (postoperative week 14).
  It will be assessed using the Fremantle Back Awareness Questionnaire.

SECONDARY OUTCOMES:
Trunk Muscle Endurance Assessment | All primary and secondary outcomes will be assessed at baseline (postoperative week 6) and post-intervention (postoperative week 14).
  The McGill Endurance Tests will measure the endurance of the trunk flexor and lateral muscles.
Lower Extremity Reaction Time Assessment | All primary and secondary outcomes will be assessed at baseline (postoperative week 6) and post-intervention (postoperative week 14).
  The motor response time to visual stimuli will be evaluated using the FITLIGHT® system.
Balance Assessment | All primary and secondary outcomes will be assessed at baseline (postoperative week 6) and post-intervention (postoperative week 14).
  Static postural control will be measured using the one-leg stance test.
Functional Performance Assessment | All primary and secondary outcomes will be assessed at baseline (postoperative week 6) and post-intervention (postoperative week 14).
  Functional mobility will be assessed using the timed up and go test.

OTHER OUTCOMES:
Level of compliance with educational recommendations | Postoperative week 6
  Participants' level of compliance with the back training and daily life recommendations provided to them during the postoperative period will be assessed using a self-report form.
Additional interventions | Up to 8 weeks
  Participants will be asked whether they are receiving any other physical therapy, exercise program, or conservative treatment, and this information will be recorded.
Adverse event and adverse reaction monitoring | Up to 8 weeks
  Any increase in pain, musculoskeletal complaints, or other potential adverse events that may occur during the exercise will be questioned and recorded during the sessions. Intervention will be terminated if necessary.
Drop-out and withdrawal reasons | Up to 8 weeks
  The reasons for participants leaving the study (lack of motivation, health issues, incompatibility, etc.) will be documented and reported in the analyses.
Adherence to exercise sessions | Post-intervention (postoperative week 14)
  The therapist will record participants' level of attendance at exercise sessions. Attendance at at least 80% of total sessions will be considered sufficient exercise compliance.
Sociodemographic and clinical characteristics | Post-operative day 1
  Gender
Sociodemographic and clinical characteristics | Post-operative day 1
  Age (years)
Sociodemographic and clinical characteristics | Post-operative day 1
  Body mass index (kg/m2)

CONTACTS AND LOCATIONS:
Overall Officials: İsmet Tümtürk, MSc, Study Chair — Süleyman Demirel University; Ferdi Başkurt, PhD, Study Director — Süleyman Demirel University; Cezmi Türk, Principal Investigator — ANTALYA PROVINCAL HEALTH DIRECTORATE ANTALYA TRAINING AND RESEARCH HOSPITAL; Fatih Özden, Principal Investigator — Muğla Sıtkı Koçman University
Locations (1):
- Antalya Provincal Health Directorate Antalya Training and Research Hospital, Antalya, Turkey (Türkiye)